CLINICAL TRIAL: NCT06443554
Title: Evaluation of the Effectiveness of a Community Health Management Program for Dry Eye Disease in Middle-Aged and Elderly Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zhang Shiyan, Director, Fujian University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ks-61-1
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Procedure: Health Management Intervention Program
- Control group (Placebo Comparator)
  Interventions: Procedure: Standard Treatment

INTERVENTIONS:
Procedure: Health Management Intervention Program — This study implemented a 12-week eye health management intervention program based on the Protection Motivation Theory (PMT). The intervention included eye health interventions conducted twice weekly at community health service locations.During the health management process, specialist doctors from higher-level comprehensive hospitals provided professional guidance, while community general practitioners took on a leading role. They provided personalized eye health management for patients under the guidance of the PMT theory. The intervention content included group education, individual guidance, experience sharing meetings, and traditional Chinese medicine appropriate technology, among other aspects.
  Arms: Intervention group
Procedure: Standard Treatment — Each week, patients were subjected to standard treatment and follow-up procedures, including basic interventions, medication, and routine follow-up via phone or WeChat, during which general conditions were assessed.
  Arms: Control group

SUMMARY:
This study evaluates the effectiveness of a community health management program for middle-aged and elderly patients with dry eye disease (DED). By comparing the community-based health management plan with conventional treatment, the study aims to determine the impact on eye health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting the diagnostic criteria for dry eye disease.
2. Middle-aged and elderly individuals aged 45 years and above.
3. Normal cognitive and expressive abilities.
4. Informed consent and ability to complete the survey.
5. Voluntary participation in the study.

Exclusion Criteria:

1. Patients with other ocular surface diseases, including stye, trachoma, allergic conjunctivitis, etc.
2. Patients with severe cataracts, glaucoma, uveitis, retinal detachment, optic nerve diseases, high myopia, or other conditions.
3. Patients who have undergone eye surgery or have a history of eye trauma in the past three months.
4. Patients who did not sign the informed consent form.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) | 12 weeks
  GAS is an individualized assessment method encompassing multiple personal goals, with a standardized formula for calculating total scores to facilitate comparisons. A score of 50 represents the expected level of achievement, with higher scores indicating greater goal attainment. GAS demonstrates good reliability, validity, and sensitivity. Based on the GAS goal list, researchers and participants collaboratively select goals and assign weights. Expected goals (assigned 0 points) and other goal levels (significantly above expected +2, slightly above expected +1, slightly below expected -1, significantly below expected -2) are established. Goal attainment is evaluated during follow-up, and GAS scores are calculated.
Ocular Surface Disease Index (OSDI) | 12 weeks
  The OSDI questionnaire assesses common dry eye symptoms and their frequency, aiding in the grading of dry eye severity. It focuses on symptoms such as dryness, foreign body sensation, stinging, photophobia, blurred vision, and the impact on daily life and environmental factors. Symptoms are rated on a scale of frequency: always (4 points), most of the time (3 points), half of the time (2 points), occasionally (1 point), and never (0 points). The OSDI total score is calculated as (sum of item scores × 25)/12, ranging from 0 to 100, with higher scores indicating more severe symptoms.
Schirmer I Test | 12 weeks
  The Schirmer I test measures tear secretion by placing a Schirmer strip under the lower eyelid conjunctiva with the patient's eyes closed, measuring tear absorption over 5 minutes. This test is widely used to evaluate dry eye syndrome. Tear secretion measured by Schirmer I test (without anesthesia) >5 mm/5 min and ≤10 mm/5 min indicates mild dry eye; >3 mm/5 min and ≤5 mm/5 min indicates moderate dry eye; and ≤3 mm/5 min indicates severe dry eye.
Quality of Life for Dry Eye Patients | 12 weeks
  NEI-VFQ-25：This is one of the most commonly used ophthalmic quality of life questionnaires, assessing vision-related issues and patients' quality of life. It consists of 25 questions divided into three parts: general health and vision, limitations in activities, and responses to vision problems. The items are categorized into dimensions such as overall health, overall vision, eye pain, near activities, distance activities, peripheral vision, color vision, driving, social functioning, role limitations, dependency, and mental health. Respondents rate their subjective experience on a 5 or 6-point scale, with scores weighted according to the question type, using values such as 100, 75, 50, 25, 0, or not scored. The highest possible score is 100, and the lowest is 0. Scores for each dimension are averaged, and overall scores for each section are averaged from the dimension scores. Higher scores indicate better quality of life.
  8.Diagnostic Criteria for Dry eye disease (DED).

CONTACTS AND LOCATIONS:
Locations (1):
- The Third People's Hospital Affiliated to Fujian University of Traditional Chinese Medicine, Fuzhou, Fujian, China